CLINICAL TRIAL: NCT04705038
Title: A Feasibility Study of Orchiectomy in Patients With Prostate Cancer on Chronic LHRH Agonist or Antagonist Therapy
Brief Title: Effect of Education on Treatment Decision Making for Patients With Prostate Cancer on Chronic Hormone Treatments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB20-0736
Record Dates: First submitted 2021-01-06; First posted 2021-01-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Intervention (Experimental): Participants in this arm undergo a short educational session about orchiectomy. They will also be asked to complete questionnaires.
  Interventions: Behavioral: Patient Education
- No Intervention (No Intervention): Participants that decline the education session will continue with routine care of their cancer.
  They will also be asked to complete questionnaires.

INTERVENTIONS:
Behavioral: Patient Education — Brief educational session on surgical castration as an alternative to lifelong ADT for prostate cancer.
  Arms: Educational Intervention

SUMMARY:
The purpose of this study is to learn how an educational intervention about orchiectomy as an alternative to medical castration for those who are already on medical castration will impact the number of patients willing to undergo an orchiectomy (surgery to remove the testicles).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic prostatic adenocarcinoma
* Receiving luteinizing hormone-releasing hormone (LHRH) agonist or LHRH antagonist therapy continuously for at least 1 year with anticipated lifelong therapy
* Able to complete written surveys in English

Exclusion Criteria:

* More than 2 prior systemic treatment regimens utilized in addition to castration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients that undergo orchiectomy after receiving study education intervention | 1 year

SECONDARY OUTCOMES:
Number of patients that agree to participate in an educational session on surgical orchiectomy | 1 year
Correlation of orchiectomy acceptance with race, socioeconomic status, level of education, and marital status. | 1 year
Change in body image perception using the Hopwood BIS questionnaire in patients undergoing versus not undergoing orchiectomy. | 1 year
Change in sexuality measured using the PROMIS v2.0 questionnaire in patients undergoing versus not undergoing orchiectomy. | 1 year
Patient satisfaction with decision to under undergo orchiectomy as reported using the Regret Decision Scale. | 1 year
  Results of patient reported satisfaction regarding their decision to undergo orchiectomy will be reported based on responses to validated Decision Regret Scale questionnaire. Higher regret scores will be associated with dissatisfaction with the decision, lower regret scores will be associated with satisfaction regarding treatment decision.
Comparison of costs of medical versus surgical castration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No